CLINICAL TRIAL: NCT07348185
Title: Clinical Evaluation of Re-treatment of Cleft Lip and Nasal Deformation in Patients With Post Repair Deformities. A Single Group Study
Brief Title: Clinical Evaluation of Re-treatment of Cleft Lip and Nasal Deformation in Patients With Post Repair Deformities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 723/2023
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Re-treatment of Cleft Lip and Nasal Deformation
Keywords: Secondary repair of Cleft Lip and Nasal Deformation; Clinical Evaluation; Cleft Q Scale; Photographic Evaluation for Lip and Nose; Radiographic assessment
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: The study was conducted after the approval of the Research Ethics Committee (REC) of the Faculty of Dentistry, Suez Canal University. It was conducted on twenty five patients who will have a secondary repair for cleft lip or nasal deformities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Twenty five patients who will have a secondary repair for cleft lip or nasal deformities. (Other): Twenty five patients who will have a secondary repair for cleft lip or nasal deformities.
  Interventions: Procedure: Procedure / Surgery

INTERVENTIONS:
Procedure: Procedure / Surgery — Procedure / Surgery

SUMMARY:
Clinical Evaluation of Re-treatment of Cleft Lip and Nasal Deformation in Patients With Post Repair Deformities. A Randomized Controlled Study

DETAILED DESCRIPTION:
Cleft lip and palate are among the most common congenital craniofacial anomalies, affecting approximately 1 in every 700 live births worldwide. These deformities can have a profound impact on both the appearance and function of the face, particularly the upper lip and nose The etiology and mode of transmission of CLP is very complex because of the congenital anomalies that are associated with it. The etiological factors include heredity, fetal environment, and environmental risk factors for CL/P such as stress, consanguinity, smoking, alcohol ingestion, use of medication during pregnancy, insufficient ingestion of folic acid in the pregestational period and in the first quarter of pregnancy, a past of miscarriage and/or stillbirth, maternal diseases, and a family history of clefts. CLP is polygenic and multifactorial involving both genetic and environmental influences.

Primary surgical repair is usually performed within the first year of life to restore anatomical continuity and function, many patients are left with residual deformities that become more apparent with growth and facial development. These secondary deformities especially involving the lip, nose, and surrounding soft tissue can significantly affect speech, feeding, dentofacial growth, and psychosocial well-being.

The secondary cleft lip and nasal deformities result from multiple factors, including scar contracture, inadequate muscle alignment, asymmetrical healing, or underlying skeletal discrepancies. The most frequently reported issues include lip tightness or shortening, irregular cupid's bow, nostril asymmetry, alar collapse, nasal septum deviation, and hypertrophic or immature scarring. Such deformities not only compromise facial aesthetics but also negatively impact the patient's psychological and social life, especially during adolescence and early adulthood.

Secondary surgical correction plays a vital role in addressing these residual issues. These procedures may include scar revision techniques such as Z-plasty or V-Y advancement, nasal tip or alar reshaping, septoplasty, cartilage grafting, fat or dermal filler injections, and lip muscle repositioning. The goal of these interventions is to restore function, achieve better symmetry, and improve the patient's overall quality of life. While the primary aim of early cleft repair is to ensure basic function and appearance, secondary interventions are often more nuanced, focusing on refinement, symmetry, and psychosocial outcomes.

Assessment of these procedures, however, must go beyond traditional clinical evaluation. Patient-reported outcome measures (PROMs) such as the CLEFT-Q have emerged as validated tools that allow the patient's voice to be integrated into outcome assessment. The CLEFT-Q assesses multiple domains including facial appearance, speech, eating, school and social functioning, and psychological well-being. It is an essential instrument for understanding the true impact of secondary cleft surgeries from the patient's perspective.

This study aimed to evaluate and manage the reconstructed cleft lip and nose deformities and secondary correction results.

The current comparative clinical study conducted at the Department of Maxillofacial Surgery Faculty of Medicine, performed on sixteen patients with Maldon cleft lip and noses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cleft lip with or without nose deformities who had undergone primary lip repair but had not yet been repaired in children and adult.

Exclusion Criteria:

* Cleft lip patients are associated with other maxillofacial congenital malformations.
* Patient, parents or care giver who did not agree to participate in the study.
* Uncooperative patients.

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
CLEFT-Q | Postoperative follow-up every week for 1 month, then after 3 and 6 months
  - The CLEFT-Q is a rigorously developed patient-reported outcome (PRO) measure that can be used internationally to collect and compare evidencebased outcomes data from patients with cleft lip and/or palate (CL/P).
  The CLEFT-Q is composed of 12 independently functioning scales and checklist.
  - Postoperative follow-up every week for 1 month, then after 3 and 6 months will be examined face, nose, nostrils, teeth, jaws, cleft, lip scar, psychological function, school function, social function speech distress, eating and drinking according to CLEFT-Q© Scales: CLEFT-Q© Scales: The CLEFT-Q© scales include number of items, ages and cleft type, recall period for completing and grade reading level.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry - Suez Canal University, Ismailia, Egypt